CLINICAL TRIAL: NCT03971435
Title: Head Start Family and Child Experiences Survey (FACES 2019)
Acronym: FACES 2019
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sara Bernstein, Principal Researcher, Mathematica Policy Research, Inc.
Other Study IDs: 50515A
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Head Start Participation
Keywords: child care; child development; child health; child nutrition; child rearing; children; curriculum; early childhood education; families; Head Start; parenting skills; parents; school readiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head Start children and families - 2019: children (2,260), parents (2,260), classrooms/teachers (590), program directors (165), center directors (318)

SUMMARY:
For over two decades, the Head Start Family and Child Experiences Survey (FACES) has been an invaluable source of information on the Head Start program and the children and families it serves. FACES 2019 extends a previously conducted data collection to a new sample of Head Start programs, families, and children. Mathematica and its partners, Juárez and Associates, Educational Testing Service, and consultants Margaret Burchinal and Martha Zaslow, developed instruments and data collection procedures to assess the school readiness skills of 2,260 children and survey their parents and Head Start teachers in fall 2019 and spring 2020 and conduct observations in Head Start classrooms and survey Head Start staff in spring 2020 and spring 2022. Due to the COVID-19 pandemic, spring 2020 child assessments and classroom observations were canceled while surveys of parents and staff continued. The pandemic and a heightened interest in the Head Start workforce brought a shift in approach and focus to spring 2022 data collection activities. As a result, those activities are not described here and instead are listed under NCT06512740.

DETAILED DESCRIPTION:
The Head Start Family and Child Experiences Survey 2019, or FACES 2019, is the seventh in a series of national studies of Head Start, with earlier studies conducted in 1997, 2000, 2003, 2006, 2009, and 2014. (FACES 2014 is entered as NCT03705377). It includes nationally representative samples of Head Start programs and centers, classrooms, children and their families. Data from surveys of Head Start program and center directors, classroom teachers, and parents provide descriptive information about program policies and practices, classroom activities, and the background and experiences of Head Start staff and families. Children in the study participate in a direct assessment that provides a rich picture of their school readiness skills at different time points.

FACES 2019 extends a previously conducted data collection to a new sample of Head Start programs, families, and children. As with previous rounds, FACES 2019 collects information from a national probability sample of Head Start programs to learn what progress Head Start has made toward meeting program performance goals.

The goals of FACES 2019 are to describe: (1) the characteristics of Head Start classrooms, programs, and staff for specific program years; (2) the changes or trends in the characteristics of classrooms, programs, and staff over time; (3) the school readiness skills and family characteristics of children who participate in Head Start during specific program years; (4) the changes or trends in children's outcomes and family characteristics over time; and (5) the factors or characteristics at multiple levels that predict differences in children's outcomes. Originally, FACES 2019 also sought to observe Head Start classroom quality but was unable to do so, with classroom observations cancelled due to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria: the Head Start programs participating in FACES 2019 were a probability sample selected from among 3,400 study-eligible programs on the 2017-2018 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be:

* In one of the 50 states or the District of Columbia
* Providing services directly to children ages 3 to 5
* The Head Start Program Performance Standards require that children turn 3 by date used to determine eligibility for public school in the community in which the Head Start program is located. Therefore, some study children were 2 years old at the time of sampling if sampling occurred before the date used for public school eligibility.
* Not be in imminent danger of losing its grantee status. Probability samples of centers were selected within each program, classrooms within each center (within those classrooms, eligible classrooms needed to have at least one Head Start child enrolled) and children within each classroom. Teachers associated with selected classrooms were included in the study with certainty, as were parents associated with selected children.

Exclusion Criteria: American Indian and Alaska Native Head Start programs (Region XI) or Migrant and Seasonal Worker Head Start programs (Region XII) were not eligible. Other ACF studies (AI/AN FACES-NCT040046965 and MSHS-NCT03116243) focus on those programs.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head Start children (and their families), Head Start programs, Head Start centers, Head Start classrooms/teachers
Sampling Method: Probability Sample
Enrollment: 5593 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
English proficiency | September to December 2019
  Children's English language proficiency were assessed during week-long site visits using Preschool Language Assessment Survey (preLAS 2000): Simon Says and Art Show. See Duncan and DeAvila for more information on the scores and technical properties.
Language-English receptive vocabulary | September to December 2019
  Indicators of language were assessed during week-long site visits using Peabody Picture Vocabulary Test-Fifth Edition (PPVT-5). See Dunn 2019 for more information on the scores and technical properties.
Language-Expressive vocabulary | September to December 2019
  Indicators of language were assessed during week-long site visits using Expressive One-Word Picture Vocabulary Test-Fourth Edition (EOWPVT-4 or EOWPVT-4 Spanish-Bilingual Edition). See Martin and Brownell 2010 and Martin 2012a for more information on the scores and technical properties.
Language-Spanish receptive vocabulary | September to December 2019
  Indicators of language were assessed during week-long site visits using Receptive One-Word Picture Vocabulary Test - Fourth Edition (Spanish-Bilingual Edition; ROWPVT-4:SBE). Please see Martin 2012b for more information on the scores and technical properties.
Literacy-Letter word knowledge | September to December 2019
  Indicators of literacy were assessed during week-long site visits using Letter-Word Identification Test from Woodcock-Johnson IV Tests of Achievement-Fourth Edition. Please see Schrank et al. 2014 and Woodcock et al. 2004 for more information on the scores and technical properties.
Literacy-early writing | September to December 2019
  Indicators of literacy were assessed during week-long site visits using Spelling Test from Woodcock-Johnson IV Tests of Achievement-Fourth Edition. Please see Schrank et al. 2014 and Woodcock et al. 2004 for more information on the scores and technical properties.
Literacy-Letter sounds knowledge | September to December 2019
  Indicators of literacy were assessed during week-long site visits using ECLS-B Letter Sounds. Please see Snow et al. 2007 for more information on the scores and technical properties
Mathematics | September to December 2019
  Indicators of mathematics were assessed during week-long site visits using the Early Childhood Longitudinal Study-Birth Cohort (ECLS-B) preschool mathematics assessment of children's understanding of relative size, ordinal numbers, and pattern matching; number recognition; and the children's ability to count, recognize shapes, add, and solve word problems. Please see Snow et al. 2007 for more information on the scores and technical properties.
Mathematics | September to December 2019
  Indicators of mathematics were assessed during week-long site visits using the Woodcock-Johnson IV Tests of Achievement-Fourth Edition/Batería III Woodcock-Muñoz (Applied Problems Test). Please see Schrank et al. 2014 and Woodcock et al. 2004 for more information on the scores and technical properties.
Children's physical health | September to December 2019
  Indicators of physical well-being were assessed by weighing (using kilograms) and measuring children's height (using centimeters), and combining these measurements to calculate Body Mass Index (BMI) in in kg/m^2.
General health status | September to December 2019
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor
Executive function | September to December 2019
  Indicators of executive function were assessed by the Minnesota Executive Function Scale (MEFS). The MEFS is a standardized and adaptive assessment administered on a touch-screen tablet with child-friendly graphics, avatars, and child-directed instructions. The MEFS provides an objective assessment of children's self-regulation, particularly cognitive flexibility, working memory, and inhibitory control. See Carlson and Zelazo 2014 for more information on the task.
Social-emotional development | September to December 2019, April-July 2020
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the FACES 2014 User's Manual (Kopack Klein et al. 2017) for more information on the scores and technical information.
Social-emotional development-cognitive/social behaviors | September to December 2019
  Indicators of social-emotional development were assessed using assessor report children's cognitive/social behaviors during the assessment time, using the Leiter International Performance Scale-Third Edition Examiner Rating Scale. The Leiter comprises eight subscales that examine children's approach to the assessments, their engagement with the materials, and their ability to attend to and regulate their physical and emotional responses during the assessment tasks. Please see Roid et al. 2013 for more information on the scores and technical properties.
Social-emotional development - Approaches to learning | September to December 2019, April-July 2020
  Indicators of social-emotional development were assessed using teacher report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
Parents' depressive symptoms | September to December 2019, March-July 2020
  Parents' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Teachers' depressive symptoms | March-July 2020
  Teachers' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bernstein, Ph.D., Study Director — Mathematica Policy Research, Inc.; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research, Inc.; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica Policy Research, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
FACES 2019 archived data are available for access.
Time Frame: Data from 2019 and 2020 are currently available.
Access Criteria: Applications for access to restricted-use data file include completing and adhering to a User Agreement.
URL: https://www.childandfamilydataarchive.org/cfda/archives/cfda/studies/38026

REFERENCES:
- [Background] Duncan, S.E., and E. DeAvila. Preschool Language Assessment Survey 2000 Examiner's Manual: English Forms C and D. Monterey, CA: CTB/McGraw-Hill, 1998.
- [Background] Dunn, D. M. Peabody Picture Vocabulary Test, Fifth Edition. Manual. Bloomington, MN: NCS Pearson, Inc., 2019.
- [Background] EOWPVT-4: Martin, N., and R. Brownell. Expressive One-Word Picture Vocabulary Test-4th Edition. Novato, CA: Academic Therapy Publications, 2010.
- [Background] EOWPVT-4:SBE: Martin, N. Expressive One-Word Picture Vocabulary Test-4th Edition: Spanish-Bilingual Edition. Novato, CA: Academic Therapy Publications, 2012.
- [Background] ROWPVT-4:SBE: Martin, N. Receptive One-Word Picture Vocabulary Test-Fourth Edition: Spanish-Bilingual Edition. Novato, CA: Academic Therapy Publications, 2012.
- [Background] Schrank, F., K. McGrew, and N. Mather. Woodcock-Johnson IV Tests of Cognitive Abilities and Achievement. Boston, MA: Houghton Mifflin Harcourt, 2014.
- [Background] Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06). NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
- [Background] Woodcock, Richard W., Ana F. Munoz-Sandoval, Kevin McGrew, Nancy Mather, and Fred Schrank. Bateria III Woodcock-Munoz. Itasca, IL: Riverside Publishing, 2004.
- [Background] Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. Reflection Sciences, Inc. St. Paul, MN.
- [Background] Kopack Klein, A., B. Lepidus Carlson, N. Aikens, A. Li, S. Bernstein, M. Dang, M. Scott, S. Skidmore, J. Cannon, N. Reid, S. Rakibullah, and L. Malone.
- [Background] Roid, G.H., L.J. Miller, M. Pomplu, and C. Koch. Leiter International Performance Scale-3rd Edition. Wood Dale, IL: Stoelting, 2013.
- [Background] U.S. Department of Education, National Center for Education Statistics. Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade. NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.
- [Background] Pianta, Robert, K. LaParo, and B. Hamre. The Classroom Assessment Scoring System Pre-K Manual. Charlottesville, VA: University of Virginia, 2008.
- [Background] Harms, T., R.M. Clifford, and D. Cryer. Early Childhood Environment Rating Scale: Revised Edition. New York: Teachers College Press, 2005.
- [Background] Clifford, Richard, Oscar Barbarin, Florence Chang, Diane M. Early, Donna Bryant, Carollee Howes, Margaret Burchinal, and Robert Pianta. What Is Pre-Kindergarten? Characteristics of Public Pre-Kindergarten Programs. Applied Developmental Science, vol. 9, no. 3, 2005, pp. 126-143.
- [Background] Kopack Klein, A., B. Lepidus Carlson, N. Aikens, A. Li, S. Bernstein, M. Dang, M. Scott, S. Skidmore, J. Cannon, N. Reid, S. Rakibullah, and L. Malone. "Head Start Family and Child Experiences Survey (2019) User's Manual." Report submitted to the Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services. Washington, DC: Mathematica, 2021.
- [Background] Radloff, L. "The CES-D Scale: A Self-Report Depression Scale for Research in the General Population." Applied Psychological Measurement, vol. 1, no. 3, 1977, pp. 385-401.
- See also: To learn more about FACES and access reports/products, please visit the FACES ACF website. — https://www.acf.hhs.gov/opre/project/head-start-family-and-child-experiences-survey-faces-1997-2022